CLINICAL TRIAL: NCT01376895
Title: Developing and Testing of an HIV Prevention Intervention Targeting Black Men Who Have Sex With Men and Women (BMSM/W)
Brief Title: Project Power: An HIV Risk Reduction Intervention for Black Men Who Have Sex With Men and Women (BMSM/W)
Acronym: Power
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: Cook County Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: POWER; 5UR6PS0011095 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Unsafe Sex; Risk Reduction
Keywords: Black MSM/W; HIV
MeSH Terms: conditions — Unsafe Sex; Risk Reduction Behavior | interventions — Advance Directives

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- POWER (Experimental): Power is a 3 session intervention delivered through the internet in real time by a trained health educator. It focuses on reducing HIV risk. Each session last from 1 to 2 hours.
  Interventions: Behavioral: PROJECT POWER
- Power Health (Active Comparator): Power Health is a 1 session general health promotion program designed to be delivered via the internet in real time by a trained health educator. The sessions focus on healthy life styles, cardiovascular health, and prostate health. Participants also receive information regarding safe sex.
  Interventions: Behavioral: Power Health

INTERVENTIONS:
Behavioral: PROJECT POWER — POWER is a three session intervention to help Black men who have sex with men and women lead healthier lives, make informed sexual choices and reduce their chances of getting or giving HIV to their sex partners. Interventions are designed to be delivered via the internet in real time by a trained health educator. Each session will last between 1 and 2 hours. The sessions are grounded on the social learning theory and use cognitive behavioral approaches. Participants learn the multiple influences on their behavior, how to identify their triggers and then use problem solving skills to develop a safer strategy for life. The sessions use videos and games to teach the lessons; participants are also given work that they must complete between the sessions.
  Arms: POWER
Behavioral: Power Health — Power Health is a one session intervention designed to help Black men who have sex with men and women improve their general health. It focuses on health issues (including HIV) that affect Black men. The program consists of 1 session delivered via the internet in real time by a trained health educator and last approximately 2 hours
  Arms: Power Health

SUMMARY:
The goal of this study is to develop and test a program to help Black men who have sex with men and women reduce their chances of getting or giving HIV infection to their sex partners. The program is designed to be delivered via the internet so that it would be available to more men. Men who agree to participate in the study will be assigned by chance to receive the POWER intervention or a similar program that is focused on general health called POWER-HEALTH. They will also complete a computer administered interview when they first enroll in the study, 2 weeks following the last session of the program and 3 months after that. Participants will receive a small compensation for their time and effort.

DETAILED DESCRIPTION:
The purpose of this study is to examine the preliminary efficacy, feasibility and acceptability of delivering a culturally and developmentally tailored HIV risk reduction intervention via the Internet in real-time that promotes risk reduction among black men who have sex with men and women (BMSMW). During the Developmental Phase, our activities will consist of completing development (finalizing sessions, completing the manuals) of a theoretically grounded, culturally based, individual intervention, Project POWER, to reduce risk of HIV acquisition and transmission among BMSMW.

The investigators will then conduct a randomized controlled trial (RCT) to test the preliminary efficacy, acceptability, and feasibility of POWER compared to HEALTH. Using chain referral methods, the investigators will recruit 200 BMSMW (100 per arm) and assign them to 1 of 2 conditions (POWER or HEALTH). Participants will complete an assessment battery delivered via ACASI at baseline, immediate post intervention and at 3 months post intervention. The investigators will also measure uptake of HIV and STI testing. Participants will also complete acceptability/feasibility assessments after the

ELIGIBILITY:
Inclusion Criteria:

* Self identify as Black or African descent
* At least 18 years of age
* Resident of Chicago MSA
* Sexually active with men and women

Exclusion Criteria:

* Previously participated in the study
* Identify as transgendered

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 211 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
unprotected sex | last 3 month
  Unprotected sex refers to either vaginal or anal sex

SECONDARY OUTCOMES:
number of sex partners | last 3 months
  number of sex partners refers to either male or female sex partners

CONTACTS AND LOCATIONS:
Locations (1):
- John H. Stroger Hospital of Cook county, Chicago, Illinois, United States